CLINICAL TRIAL: NCT07216131
Title: A Fixed-sequence, Open-label Study to Assess the Effect of AZD0780 on the Pharmacokinetics of Metformin in Healthy Volunteers
Brief Title: A Study to Investigate the Effect of AZD0780 on Metformin Pharmacokinetics in Healthy Adult Volunteers Aged 18 to 55 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7960C00003
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Renal Transporter; Multidrug and Toxic Compound Extrusion 1; Dyslipidemia; Proprotein Convertase Subtilisin/Kexin Type 9
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin/Metformin + AZD0780 (Experimental): Participants will receive a single dose of metformin on Day 1 in Treatment Period 1 followed by a washout period of 7 days. In Treatment Period 2, participants will receive a single dose of AZD0780 followed by a single dose of metformin on Day 8.
  Interventions: Drug: AZD0780; Drug: Metformin

INTERVENTIONS:
Drug: AZD0780 — AZD0780 will be administered orally.
Drug: Metformin — Metformin will be administered orally.

SUMMARY:
The purpose of this study is to determine how the experimental medication AZD0780 impacts the pharmacokinetics (PK) of metformin, a common medication used to treat type 2 diabetes mellitus, when given together in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, 2-period, fixed-sequence study in healthy participants (males and females), performed at a single Clinical Unit. The study will assess the PK of metformin when administered alone and in combination with a single dose of AZD0780.

The study will comprise:

* A Screening Period of maximum 28 days.
* Two Treatment Periods (Day -1 to Day 7 and Day 8 to Day 10) during which participants will be resident at the Clinical Unit and will receive the study intervention.
* A final Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 35 kilograms per meter squared (kg/m2) inclusive and weigh at least 50 kilograms (kg) at the Screening Visit.
* Participants agree to follow study specific contraceptive requirements.
* Have suitable veins for cannulation or repeated venipuncture.

Exclusion Criteria:

* History of any clinically important disease or disorder which may put the participant at risk because of participation in the study or influence the results.
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to metformin or AZD0780.
* Treatment with any lipid lowering therapy or AZD0780 within the 3 months prior to the Screening Visit.
* Treatment with drugs for reduction or inhibition of proprotein convertase subtilisin/kexin type 9 (PCSK9) within the last 12 months prior to the Screening Visit (approved or investigational and apart from AZD0780).
* Current or previous administration of inclisiran.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-11-10 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on the PK of metformin.
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on the PK of metformin.
Maximum observed drug concentration (Cmax) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on the PK of metformin.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Day 1 until Follow-up visit or early discontinuation (Up to Day 18)
  To examine the safety and tolerability of AZD0780 in combination with metformin.
Apparent total body clearance (CL/F) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Apparent volume of distribution based on the terminal phase (Vz/F) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Terminal elimination half life (t½λz) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Time to reach maximum observed concentration (tmax) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Renal clearance (CLR) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Amount of unchanged drug excreted into urine (Ae) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.
Percentage of dose excreted unchanged in urine (fe) | Days 1 to 3 and Days 8 to 10
  To assess the effect of AZD0780 on other PK parameters of metformin.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. ''Yes", indicates that AZ is accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Thank You Card — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00003&attachmentIdentifier=847613b1-21d0-4b0c-8a52-389ac3ab70c9&fileName=AZ_D7960C00003_TY_v1.0_2025_09_23_-_Finalized.pdf&versionIdentifier=